CLINICAL TRIAL: NCT06007014
Title: A Multi-Center, Randomised, Double-blind, Placebo Parallel Controlled Clinical Study to Evaluate the Efficacy and Safety of Chiglitazar Added to Glargine in Patients With Type 2 Diabetes
Brief Title: Efficacy and Safety of Chiglitazar Added to Glargine in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanbing Li (Other)
Responsible Party: Sponsor-Investigator, Yanbing Li, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLi
Record Dates: First submitted 2023-07-26; First posted 2023-08-23 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Efficacy and Safety of Chiglitazar Sodium in the Treatment of T2DM Patients; Metformin Combined With Insulin Glargine in the Treatment of Type 2 Diabetes Patients Who Still Have Poor Hypoglycemic Effect; 128 Patients Were Randomly Assigned 1:1; Metformin and Insulin Glargine Combined With Chiglitazar Sodium Tablets 48mg/ Day Group; Metformin and Insulin Glargine Combined With Placebo Group; InvestigatorInitiate Trial; Changes in HbA1C From Baseline at 18 Weeks of Treatment
Keywords: Chiglitazar; T2DM; Randomised; Double-blind; Placebo Parallel Controlled

STUDY DESIGN:
Intervention Model Description: Metformin and insulin glargine combined with Chiglitazar sodium tablets 48mg/ day group；Metformin and insulin glargine combined with placebo group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Metformin and insulin glargine combined with sitaglitat sodium tablets 48mg/ day group;
  Interventions: Drug: Chiglitazar sodium
- Placebo group (Placebo Comparator): Metformin and insulin glargine combined with placebo group
  Interventions: Drug: Chiglitazar placebo

INTERVENTIONS:
Drug: Chiglitazar sodium — tablets 48mg/ day administered for 18 weeks
  Arms: Intervention group
Drug: Chiglitazar placebo — tablets 48mg/ day administered for 18 weeks
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to evaluate the Efficacy and Safety of Chiglitazar Added to Patients with type 2 diabetes who do not respond well to metformin combined with insulin glargine. The main question it aims to answer are:

• T2DM patients still cannot effectively control their blood sugar with the combination of insulin and metformin. The combination of follow-up treatment and hypoglycemic drugs is worth exploring, and it is necessary to explore and confirm the combination of effective and safe drugs for insulin resistance on the basis of the above treatment plans.

Participants will be asked to receive either Chiglitazar or placebo in addition to metformin and insulin glargine 18 weeks.

Researchers will compare placebo groups to see if the effective effect and safety indicators of Chiglitazar for reducing insulin dosage, lowering blood sugar, regulating blood lipids.

DETAILED DESCRIPTION:
T2DM patients using insulin combined with metformin dual therapy regimen, still can not have effective control of blood sugar, the combination of follow-up treatment and hypoglycemic drugs is worth exploring, and it is necessary to base on the above treatment plans to explore and confirm the treatment of effective and safe drugs for insulin resistance. This study investigated the efficacy and safety of metformin combined with insulin glargine in the treatment of type 2 diabetes mellitus (T2DM) in patients who still have poor hypoglycemic effect, plus Chiglitazar 48mg/ day for 18 weeks.

A total of 128 patients were expected to be included, and were randomly assigned 1:1 to the combination of metformin and insulin glargine combined with Chiglitazar sodium tablet 48mg/ day group. Metformin and insulin glargine combined with placebo group.

ELIGIBILITY:
Inclusion Criteria:

* 1.In accordance with the World Health Organization (WHO) issued in 1999 diabetes diagnostic criteriaType 2 diabetes mellitus (T2DM);
* 2. Male or female patients ≥18 years old;
* 3, BMI≥18.5 Kg/m2, < 35 Kg/m2;
* 4, Glycosylated hemoglobin (HbA1C) > 7.5%; ≤10.5%;
* 5, Stable dose (insulin daily therapeutic dose change within ±20%) of glycerine or DI The therapeutic dose of Terterigu or NPH basal insulin is ≥0.25IU/kg/ day/or 20IU/ day；
* 6, Stable basic insulin treatment combined with metformin (metformin dose ≥1000mg/Days or maximum tolerated dose) ≥3 months；
* 7. Voluntarily sign informed consent and agree to be randomly assigned to any experimental group.

Exclusion Criteria:

* 1, Type 1 diabetes or specific type diabetes;
* 2. Fasting blood glucose (FPG) exceeding 13.3 mmol/L (240 mg/dL);
* 3, refractory hypertension [that is, on the basis of improving lifestyle, the application of a reasonable and tolerable sufficient amount of 3 or more antihypertensive drugs (including diuretics) for more than 1 month still does not reach the standard, or take 4 or more antihypertensive drugs to effectively control blood pressure];
* 4. Triglyceride (TG) > 500 mg /dL (5.65 mmol/L);
* 5, is taking or in the last 1 month has taken fibrate drug treatment;
* 6, lower limb edema or general edema;
* 7. Experienced 3 or more episodes of severe hypoglycemia and/or unintentional hypoglycemia in the 6 months prior to screening;
* 8. A definite diagnosis of osteoporosis or any other known bone disease;
* 9. History of diabetic ketoacidosis, diabetic hyperglycemia hyperosmolar syndrome, lactic acidosis and other acute complications of diabetes;
* 10. Severe microvascular complications (proliferative retinopathy; Urinary albumin/creatinine ratio > 300 mg/g; Marked peripheral neuropathy, etc.);
* 11. Large vascular lesions leading to hospital admission within 6 months before inclusion;
* 12, The New York Heart Association (NYHA) defines congestive heart failure as grade III or IV
* 13, significant liver and kidney dysfunction and systemic disease (significant liver dysfunction is defined as AST> 2.5 times the upper limit of normal and/or ALT> 2.5 times the upper limit of normal and/or total bilirubin > 1.5 times the upper limit of normal value; Renal dysfunction was defined as moderate to severe renal insufficiency (eGFR<60 ml/ (min*1.73m2)).
* 14. Use of other hypoglycemic agents not specified in the inclusion criteria (thiazolidinediones, GLP-1RA, premixed or fast-acting insulin) in the current or 3 months prior to screening, with the exception of short-term treatment with additional insulin (a total of 7 days or less) for complications;
* 15, pregnant or lactating women, women of childbearing age who are unable or unwilling to take adequate contraception;
* 16. Participating in clinical trials of other drugs or medical devices during or within 3 months prior to screening;
* 17. The investigator considers it inappropriate to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
HbA1C | 18 weeks of treatment
  Changes in HbA1C from baseline

SECONDARY OUTCOMES:
Insulin | 6 weeks and 18 weeks of treatment
  Changes in the daily dose of insulin from baseline
Triglyceride | 18 weeks of treatment
  Changes in the daily dose of triglyceride from baseline
Fasting blood glucose | 6 weeks and 18 weeks of treatment
  Changes in the daily dose of fasting blood glucose from baseline
Fasting C-Peptide | 18 weeks of treatment
  Changes in the daily dose of fasting C-Peptide from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China